CLINICAL TRIAL: NCT05512221
Title: Optimizing Engagement and Reach of a Transdiagnostic Group Therapy for Autistic Adults Through Technology and Personalized Therapeutics
Brief Title: Transdiagnostic Group Therapy (GBAT) for Autistic Adults With Personalized Therapeutics
Acronym: (GBAT+)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: New Jersey Governor's Council for Medical Research and Treatment of Autism (Unknown)
Responsible Party: Principal Investigator, Vanessa H. Bal, PhD, Associate Professor; Karmazin and Lillard Chair in Adult Autism, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022001343
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: GBAT+Individual; GBAT+Engagement Booster; GBAT+Both
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I (Experimental): GBAT+I and GBAT+E groups
  Interventions: Other: GBAT+I, GBAT+E - Phase I
- Phase 2a (Experimental): Watchful Waiting, GBAT+I, and GBAT+E groups
  Interventions: Other: Watchful Waiting and Groups - Phase 2
- Phase 2b (Experimental): GBAT+IE groups
  Interventions: Other: GBAT+IE

INTERVENTIONS:
Other: GBAT+I, GBAT+E - Phase I — Phase I is the development phase, which is informed by the study team's previous pilot study and autistic advisors. It will include the development of engagement booster materials. Booster materials will be tested in 2 groups (GBAT+I and GBAT+E) of six participants each. Groups include GBAT+Individual (GBAT+I; individual sessions to supplement the 10 group sessions) and GBAT+Engagement Booster (GBAT+E; supplemental materials). The first 4-6 eligible adults recruited will participate in GBAT+I and the second 6 eligible adults recruited will participate in GBAT+E. Both groups will consist of 10 weekly 60-90-minute GBAT group sessions. Participants in the GBAT+I group will also attend 30-minute individual booster sessions, approximately between Weeks 4-5, 5-6, 6-7, and 7-8. Participants in the GBAT+E group will be asked to use booster materials in between group sessions (e.g., worksheets, goal trackers, interactive learning activities).
  Arms: Phase I
Other: Watchful Waiting and Groups - Phase 2 — Phase 2a will include a watchful waiting (WW) condition and assignment to 1 of 2 treatment conditions: GBAT+I or GBAT+E.
  Participants will be assigned to WW for 10 wks. They will not receive specific therapeutic services during WW, but a member of the study team will contact them at weeks 1, 2, 4, 6, and 8 to maintain engagement and monitor for clinical deterioration.
  After WW, participants will be randomly assigned to one of the treatment conditions (GBAT+I or GBAT+E). All groups will consist of 10 weekly 60-90-minute GBAT group sessions. GBAT+I participants will attend four 30-minute individual booster sessions. GBAT+E participants will be asked to use booster materials between group sessions (e.g., worksheets, goal trackers, interactive learning activities)
  WW group size is based on study feasibility and availability of resources. Additional participants will also be recruited at the end of the WW period to supplement group sizes.
  Arms: Phase 2a
Other: GBAT+IE — Phase 2b will include assignment to GBAT+IE, which includes components of both GBAT+I (individual sessions) and GBAT+E (supplemental materials)
  All groups will consist of 10 weekly 60-90-minute GBAT group sessions. Participants in the GBAT+I group will also attend 30-minute individual booster sessions, approximately between Weeks 4-5, 5-6, 6-7, and 7-8. Participants in the GBAT+E group will be asked to use booster materials in between group sessions (e.g., worksheets, goal trackers, interactive learning activities). Participants in GBAT+IE will participate in both the individual sessions and use of booster materials.
  Arms: Phase 2b

SUMMARY:
The purpose of this study is to build upon an earlier study that evaluated the use of a 10-week transdiagnostic Group Behavioral Activation Therapy (GBAT), a telehealth delivered intervention, as a cost effective and accessible way to treat symptoms of anxiety and depression in autistic adults. The current study will pilot and compare relative feasibility, acceptability, and preliminary efficacy of three adapted GBAT groups and a Watchful Waiting (WW) group. The three groups include GBAT+Individual (GBAT+I; individual sessions to supplement the 10 group sessions), GBAT+Engagement Booster (GBAT+E; supplemental materials), and GBAT+Both (GBAT+IE individual sessions and supplemental materials).

ELIGIBILITY:
Inclusion Criteria:

* Live in New Jersey or New York
* Be 18-40 years old
* Have a confirmed diagnosis of Autism Spectrum Disorders (ASD).
* Have access to a device (e.g., computer with a webcam or smartphone) in order to complete online surveys and participate in videoconference sessions
* WRAT Reading Comprehension grade equivalent 6th grade or higher
* Receive a best-estimate diagnosis of an anxiety or mood disorder (Generalized Anxiety Disorder, Social Anxiety Disorder, Specific Phobia, Panic Disorder, Agoraphobia, Major Depressive Disorder, Unspecified Depression, Persistent Depressive Disorder).
* Be interested in participating in an online telehealth treatment group to address their difficulties in the aforementioned areas
* Approximately 60% of our sample will be White, Non-Hispanic; approximately 40% of our sample will be female-identifying and 40% will be male-identifying

Exclusion Criteria:

* Are younger than 18 years old, or older than 40 years old
* Do not have an ASD diagnosis
* Have WRAT Reading Comprehension below 6th grade level
* Are unable to understand English fluently
* Have a principal DSM-5 disorder other than one of the above listed anxiety or depression disorders, have received a diagnosis of Intellectual Disability, schizophrenia, or bipolar disorder or demonstrate suicidal ideation or intent severe enough to require current hospitalization, or who have attempted suicide in the past 3 months.
* Are currently enrolled in another behavioral therapy or psychotherapy targeting depression, anxiety or anger.
* Are experiencing suicidal ideation that requires current hospitalization.
* The PI's best clinical judgment that it would not be in the adult's best interest to be enrolled (e.g., due to factors that may affect their engagement or comfort in the group).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Global Impression Severity (CGIS) Scale: Independent Evaluator | Change from pre-treatment to post-treatment (an average of 12 weeks)
  The CGI-S score provides a global rating of baseline severity ranging from 1 (not at all ill) to 7 (extremely ill), while the CGI-I provides a global rating of clinical improvement ranging from 1 (Very Much Improved) to 7 (Very Much Worse). The IE will provide a baseline CGI ratings for each patient at pretreatment and posttreatment.

SECONDARY OUTCOMES:
Change in distress on Patient Health Questionnaire (PHQ-9) | Change from pre-treatment to post-treatment (an average of 12 weeks)
  The PHQ-9 is a 9-item questionnaire of psychological function over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Total scores range from 0 to 27; higher scores reflect greater levels of depressive symptoms.
Change in anxiety symptoms on the Generalized Anxiety Disorder Questionnaire (GAD-7) | Change from pre-treatment to post-treatment (an average of 12 weeks)
  The GAD-7, assessed weekly, is a 7-item questionnaire of anxiety symptoms over the past week with all items on a "0" (not at all) to "3"(nearly every day) scale. Total scores range from 0 to 21; higher scores reflect greater levels of anxiety.
Anxiety Disorders Interview Schedule for DSM-5 | Change in CSR from pre-treatment to post-treatment (an average of 12 weeks)
  The ADIS-5 is a semi-structured diagnostic interview that assesses mood and anxiety disorders. The interview focuses on clinical threshold of symptoms to inform current diagnostic presentations. Clinician Severity Rating (CSR) is rated for each diagnosis to quantify the interference of symptoms on a scale from 0 ("not at all") to 8 ("debilitating"). A score of 4 and above denotes a clinical threshold.
Behavior Rating Inventory of Executive Function - Adult Form | Change from pre-treatment to post-treatment (an average of 12 weeks)
  The BRIEF is a standardized measure that captures executive functions or self-regulation in an everyday environment. The BRIEF is composed of 75 items within nine theoretically and empirically derived clinical scales that measure various aspects of executive functioning. These scales form a Behavioral Regulation Index and Metacognition Index, as well as an overall Global Executive Composite Each of the scales and indexes yields standardized scores that allow for comparison with adults of the same age and gender (T-scores with a mean of 50 and a standard deviation of 10). T-scores between 60 and 64 are considered "Mildly Elevated," while scores between 65 and 69 are considered "Potentially Clinically Elevated." T-scores above 70 are considered "Clinically Elevated" and may warrant clinical attention.
Mirror Tracing Persistence Task | Change from pre-treatment to post-treatment (an average of 12 weeks)
  The MTPT is a behavioral task that evaluates persistence. The participant is asked to trace the outline of 3 stars (rated easy, medium, and difficult), one at a time. The thickness of each subsequent star's outline gets smaller, making it harder to trace. To increase distress, the cursor is programmed to operate in the opposite direction of the user's input. If the participant goes outside the outline, a buzzer sounds and puts the participant back at the start point. Prior to tracing any stars, the participant's affect is assessed using a 100-point scale (0 = none and 100 = extreme) to assess frustration, anxiety, happiness, irritability, difficulty concentrating, and physical discomfort. The participant traces the "difficult" star again, only this time they are given an option to quit. The participant's time is recorded to measure how long they persist on the final star, referred to as task persistence. Afterwards, they rate affect from 0-100 in order to assess change in affect.
Distress Tolerance Test | Change from pre-treatment to post-treatment (an average of 12 weeks)
  The DTT is a behavioral task that evaluates an individual's willingness to persist at a task in spite of heightened frustration and distress. It uses the stimulus cards from the Wisconsin Card Sort Test. The DTT provides consistently negative feedback over a small number of trials (thus serving as a more "compact" distress induction) and by including the opportunity to escape after 20 trials, which provides a behavioral measure of distress tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Bal, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No